CLINICAL TRIAL: NCT02728193
Title: The Research on Standard Treatments of Very-early Stage Hepatocellular Carcinoma: a Randomized Clinical Trial
Brief Title: Standard Treatments of Very-early Stage Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012ZX10002016003001
Record Dates: First submitted 2016-03-28; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; Very-early Stage
Keywords: treatments; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RFA (Experimental): Radiofrequency ablation
  Interventions: Procedure: RFA
- MWV (Experimental): Microwave ablation
  Interventions: Procedure: MWV
- PEI (Experimental): Percutaneous ethanol injection
  Interventions: Procedure: PEI

INTERVENTIONS:
Procedure: RFA
  Arms: RFA
Procedure: MWV
  Other Names: Microwave ablation
  Arms: MWV
Procedure: PEI — Percutaneous ethanol injection
  Arms: PEI

SUMMARY:
The aim of our study was to elucidate the difference in the rates of complication, hospitalization days, medical expenses, MRI showed that the degree of tumor necrosis, and overall survival rates of the therapies between PEI, MVA and RFA, and make the standard for minimally invasive treatment of very early stage HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative clinical, imaging and tumor markers were diagnosed as hepatocellular carcinoma
2. Tumor diameter<2cm
3. Child-Pugh class A liver function
4. Without major organ dysfunction
5. male or female patients > 18 years and <=70 years of age
6. Voluntary participation in this clinical trial

Exclusion Criteria:

1. Other anticancer treatment before therapy
2. Patients with apparent major organs (i.e. cardiac, pulmonary, cerebral and renal) dysfunction, which may affect the treatment of liver cancer
3. Patients with other diseases that may affect the treatment of this treatment
4. History of other malignant tumors
5. Patients who are participating in other clinical trials
6. Pregnant, lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recurrence | 3 years
  Hepatocellular Carcinoma will recurrence in 3 years
Death | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China